CLINICAL TRIAL: NCT02554929
Title: Efficacy of a Group Cognitive Behavioral Therapy Program in the Treatment of Young Children With Social Anxiety Disorder and/or Selective Mutism: A Randomized Controlled Trial
Brief Title: Treatment of Social Anxiety Disorder and Selective Mutism
Acronym: SAD&SMTRMT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Suneeta Monga, Medical Director, Psychiatry Ambulatory Services, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1000050447
Record Dates: First submitted 2015-09-15; First posted 2015-09-18 (Estimated); Results first posted 2019-09-13 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Social Anxiety Disorder; Selective Mutism
Keywords: Social Anxiety Disorder; Selective Mutism; CBT; preschool anxiety disorders
MeSH Terms: conditions — Phobia, Social; Mutism | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Taming Sneaky Fears Group (Experimental): An 11 week (introduction plus 10 week) manualized treatment protocol utilizing cognitive behavioral strategies specifically developed for children 4 to 7 years of age with social anxiety disorder and/or selective mutism. Parent and child groups run separately but concurrently.
  Interventions: Behavioral: Taming Sneaky Fears
- Parent Psychoeducation and Child Socialization Group (Active Comparator): An 11 week (introduction plus 10 week) manualized treatment protocol focusing on parent psychoeducation and child socialization in children 4 to 7 years of age with social anxiety disorder and/or selective mutism. Parent and child groups run separately but concurrently.
  Interventions: Behavioral: Parent Psycho-education and Child Socialization

INTERVENTIONS:
Behavioral: Taming Sneaky Fears — Parents receive coping strategies based on CBT in parent group and children receive coping strategies based on CBT in child group.
  Other Names: Cognitive Behavioral Therapy (CBT)
  Arms: Taming Sneaky Fears Group
Behavioral: Parent Psycho-education and Child Socialization — Parents receive psycho-education in parent group and children receive socialization skills in child group.
  Other Names: Psycho-education and Socialization
  Arms: Parent Psychoeducation and Child Socialization Group

SUMMARY:
This study is to assess the efficacy of a brief, 11-week, manualized Taming Sneaky Fears for Social Anxiety Disorder (SAD) and/or Selective Mutism (SM) child and parent group Cognitive Behavioural Therapy (CBT) treatment protocol. Children 4 to 7 years old (n = 88) meeting criteria for SAD and/or SM, and their parents are recruited from the Psychiatry Outpatient Program and participants will be randomized to either the Taming Sneaky Fears group or a parent psycho-education and child socialization group. Trained clinicians blinded to all measures and treatment assignment will administer pre, post and 6-month follow-up outcome measures. Investigators assess within-the-child and within-the-parent/environment factors that predict treatment outcomes.

DETAILED DESCRIPTION:
This study utilizes a repeated measures, longitudinal, randomized controlled trial design to compare the efficacy of two interventions in the treatment of children aged 4 to 7 years with SM and/or SAD. Participants are randomized into either the:

1. Taming Sneaky Fears for SAD and/or SM parent and child group CBT treatment, or
2. the Parent Psycho-education and Child Socialization comparison program.

Both programs run for 10 consecutive weeks (plus one additional introduction week). To control for the nonspecific factors associated with treatment, such as the support, attention and expectation of improvement, parents and children in both treatment protocols receive comparable levels of attention from therapists (i.e., same duration of group sessions and total number of sessions with a therapist) and comparable opportunities for socialization (e.g., for the children: invitation to discuss how the previous week went, snack time, story time; for the parents: discussion of specific topics at each session). However, parents and children in the comparison group are not taught CBT strategies.

ELIGIBILITY:
Inclusion Criteria:

* 4 to 7 year old children who meet diagnostic criteria for a primary diagnosis of Selective Mutism (SM) and/or Social Anxiety Disorder (SAD) through a clinical and semi-structured diagnostic interview .
* Presence of other anxiety disorders/symptoms is not an exclusion criterion as long as the main concern (primary diagnosis) is SAD and/or SM.

Exclusion Criteria:

* Presence of autism spectrum disorder, brain injury, or significant developmental delays (based on medical history and clinical assessment).
* Children and parents not fluent in English.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suneeta Monga, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Albano, A. M., & Silverman, W. K. (1996). Anxiety Disorders Interview Schedule for DSM-IV-Child Version: Clinician Manual. Psychological Corporation.
- [Background] Shaffer D, Gould MS, Brasic J, Ambrosini P, Fisher P, Bird H, Aluwahlia S. A children's global assessment scale (CGAS). Arch Gen Psychiatry. 1983 Nov;40(11):1228-31. doi: 10.1001/archpsyc.1983.01790100074010. PMID 6639293
- [Background] Bergman RL, Keller ML, Piacentini J, Bergman AJ. The development and psychometric properties of the selective mutism questionnaire. J Clin Child Adolesc Psychol. 2008 Apr;37(2):456-64. doi: 10.1080/15374410801955805. PMID 18470781
- [Background] Spence, S. H., & Rapee, R. (1999). Preschool anxiety scale (parent report). Brisbane, Australia: University of Queensland.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at the Hospital for Sick Children (SickKids). Children, aged 4-7 years, were screened to participate in the treatment study by one of the principal investigators (child psychiatrists) at an anxiety disorders clinic in SickKids.
Pre-assignment Details: Of the n=93 consented participants, 3 withdrew consent prior to randomization and treatment assignment.
Groups:
- Taming Sneaky Fears Group: An 11 week (introduction plus 10 week) manualized treatment protocol utilizing cognitive behavioral therapy (CBT) strategies specifically developed for children 4 to 7 years of age with social anxiety disorder (SAD) and/or selective mutism (SM). Parent and child groups were conducted separately but concurrently.
  Taming Sneaky Fears: Parents received coping strategies based on CBT in parent group and children received coping strategies based on CBT in child group.
- Parent Psychoeducation and Child Socialization Group: An 11 week (introduction plus 10 week) manualized treatment protocol focusing on parent psychoeducation and child socialization in children 4 to 7 years of age with social anxiety disorder (SAD) and/or selective mutism (SM). Parent and child groups were conducted separately but concurrently.
  Parent Psycho-education and Child Socialization: Parents received psycho-education in parent group and children received socialization skills in child group.
Period: Overall Study
Arm/Group | Taming Sneaky Fears Group | Parent Psychoeducation and Child Socialization Group
Started | 46 | 44
Per Protocol Received Intervention | 44 | 36
Per Protocol Post-Intervention | 42 | 36
Per Protocol 6 Month Follow-up | 40 | 32
Completed | 40 | 32
Not Completed | 6 | 12
Not completed — Lost to Follow-up | 4 | 4
Not completed — Withdrawal by Subject | 2 | 8

BASELINE CHARACTERISTICS:
Population: 4 to 7 year old children referred for psychiatric assessment of SM and/or social anxiety disorder (SAD) who met diagnostic criteria for SM and/or SAD as a primary diagnosis, as determined by one of the psychiatrists at the site where the study was conducted.
Groups:
- Total: Total of all reporting groups
Arm/Group | Taming Sneaky Fears Group | Parent Psychoeducation and Child Socialization Group | Total
Number analyzed (Participants) | 46 | 44 | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 46 | 44 | 90
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.9 (1.0) | 5.8 (1.1) | 5.9 (1.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 31 | 63
  Male | 14 | 13 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 45 | 42 | 87
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 10 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 25 | 30 | 55
  More than one race | 8 | 2 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 46 | 44 | 90
The Anxiety Disorders Interview Schedule (ADIS), Clinical Severity Rating (ADIS-CSR) [Mean (Standard Deviation); unit: units on a scale] — The ADIS-CSR was used to assess SAD and/or SM. This measure has good reliability, is sensitive to treatment effects in child anxiety studies, and has been used in a number of studies on preschoolers and SM treatment. Clinical Severity Rating (ADIS-CSR) uses a 0 to 8 scale to measure clinical severity of diagnosis; a CSR of ≥4 indicates clinically significant symptoms and presence of an anxiety disorder. A trained independent clinician blinded to treatment type and time of assessment completed the CSR.
  units on a scale
    SAD ADIS-CSR Score | 5.2 (1.7) | 5.7 (1.3) | 5.5 (1.6)
    SM ADIS-CSR Score | 4.8 (2.4) | 4.3 (2.5) | 4.5 (2.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinical Severity Ratings (CSR) of SAD & SM on the Anxiety Disorders Interview Schedule - Parent Version (ADIS-P)
Description: The Anxiety Disorders Interview Schedule for Diagnostic and Statistical Manual of Mental Disorders (DSM-IV): Parent Version (ADIS-P) is a semi-structured, clinician-administered, interview of parents used to diagnose anxiety and other related disorders in children and adolescents. Parents were asked to rate for interference or impairment using a 9-point scale ranging from 0 to 8, with 0 being not impaired or not interfering and 8 being significant impairment or interference. A final Clinician Severity Rating (CSR) was then established using the same scale, with a CSR of 4 (moderate degree of impairment) or greater required to establish a diagnosis.
Time Frame: Change from Baseline in CSR of SAD & SM at 6 months after treatment ends. Treatment groups run for 11 weeks.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Taming Sneaky Fears Group | Parent Psychoeducation and Child Socialization Group
Number analyzed (Participants) | 46 | 44
units on a scale
  Change in SAD ADIS-CSR from baseline to 6 months | -1.26 (0.35) | -1.65 (0.37)
  Change in SM ADIS-CSR from baseline to 6 months | -1.51 (0.37) | -1.24 (0.40)
Statistical Analysis 1: Comparison: Taming Sneaky Fears Group vs Parent Psychoeducation and Child Socialization Group; In our previous study, 42% participants in the CBT arm lost their primary diagnosis of social anxiety disorder (SAD) and/or selective mutism (SM) post-intervention versus none of the comparison group participants. In the present study, we conservatively estimated that 10% of comparison group children will lose their primary diagnosis. A sample size of 70 achieves a power of 81% to detect a 32% difference between treatments, using a two-sided Chi-squared test with a significance level of 0.05; Test type: Superiority; p = 0.002, Mixed Models Analysis — P value adjusted for multiple comparison; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.91 to 0.74], Standard Error of Mean 0.42 — Values above are for the primary outcome measure of the Anxiety Disorders Interview Schedule for DSM-IV, Clinical Severity Rating (ADIS-CSR) score for SAD
Statistical Analysis 2: Comparison: Taming Sneaky Fears Group vs Parent Psychoeducation and Child Socialization Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.002, Mixed Models Analysis — P value adjusted for multiple comparison; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = 0.27, 95% CI 2-sided [-0.95 to 1.48], Standard Error of Mean 0.62 — Values above are for the primary outcome measure of the Anxiety Disorders Interview Schedule for DSM-IV, Clinical Severity Rating (ADIS-CSR) score for SM

2. Secondary Outcome: Change in Clinical Severity Ratings (CSR) of SAD & SM on the Anxiety Disorders Interview Schedule - Parent Version (ADIS-P)
Description: The Anxiety Disorders Interview Schedule for DSM-IV: Parent Version (ADIS-P) is a semi-structured, clinician-administered, interview of parents used to diagnose anxiety and other related disorders in children and adolescents. Parents were asked to rate for interference or impairment using a 9-point scale ranging from 0 to 8, with 0 being not impaired or not interfering and 8 being significant impairment or interference. A final Clinician Severity Rating (CSR) was then established using the same scale, with a CSR of 4 (moderate degree of impairment) or greater required to establish a diagnosis.
Time Frame: Change from Baseline in CSR within 4 weeks of treatment end. Treatment groups run for 11 weeks.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Taming Sneaky Fears Group | Parent Psychoeducation and Child Socialization Group
Number analyzed (Participants) | 46 | 44
units on a scale
  Change in SAD ADIS-CSR baseline to 4-weeks | -1.12 (0.34) | -1.46 (0.37)
  Change in SM ADIS-CSR baseline to 4-weeks | -1.49 (0.37) | -0.66 (0.40)

3. Secondary Outcome: Change in Children's Global Assessment Scale (CGAS)
Description: The Children's Global Assessment Scale (CGAS) is a clinician rating of overall adaptive functioning during the previous month for children and adolescents between 4 to 16 years of age. CGAS scores are rated on a 100-point scale, with 1 being the most impaired and 100 being least impaired, and descriptors for each 10-point interval such that each 10-point interval defines a range of children's functioning in all areas of their life. CGAS scores were secondary outcome measures. The Change in Children's Global Assessment Scale (CGAS) measures level of general functioning on a 100 point scale - 1 (needs constant supervision) to 100 (superior functioning). Every 10 points global functioning moves to the next category.
Time Frame: Change from Baseline on the CGAS within 4 weeks of treatment end. Treatment groups run for 11 weeks.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Taming Sneaky Fears Group | Parent Psychoeducation and Child Socialization Group
Number analyzed (Participants) | 46 | 44
units on a scale | 12.8 (2.4) | 11.1 (2.5)

4. Secondary Outcome: Change in Children's Global Assessment Scale (CGAS)
Description: as for outcome 3
Time Frame: Change from Baseline on the CGAS at 6 months post-treatment end. Treatment groups run for 11 weeks.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Taming Sneaky Fears Group | Parent Psychoeducation and Child Socialization Group
Number analyzed (Participants) | 46 | 44
units on a scale | 15.2 (2.5) | 14.3 (2.6)
Statistical Analysis 1: Comparison: Taming Sneaky Fears Group vs Parent Psychoeducation and Child Socialization Group; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.002, Mixed Models Analysis — P value adjusted for multiple comparison; a priori threshold for statistical significance was 0.05; Mean Difference (Final Values) = 1.89, 95% CI 2-sided [-4.28 to 8.08], Standard Error of Mean 3.14 — The estimated value of the estimation parameter corresponds to the difference between change in CGAS scores for participants in the CBT arm, in comparison to those in the socialization arm, from pre-treatment to 6-month follow-up

5. Secondary Outcome: Selective Mutism Questionnaire (SMQ)
Description: The Selective Mutism Questionnaire (SMQ) is a 17-item parent questionnaire that assesses the degree and frequency of speech in 3-to-11-year-old children and provides a proxy measure of selective mutism severity. Parents report on their child's behavior with regards to speaking in the previous two weeks across three broad domains (or subscales): at school (five items), at home/with family (five items), and in social situations (seven items). Parents rate items using a three-point scale that ranges from 0 = never to 3 = always. Lower total scores on the Selective Mutism Questionnaire suggest less speech.
Time Frame: The SMQ was completed by parents at all 3 time-points: 1) Pre-treatment (baseline), 2) Post-treatment, and 3) 6-month follow-up (from baseline date).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taming Sneaky Fears Group | Parent Psychoeducation and Child Socialization Group
Number analyzed (Participants) | 46 | 44
units on a scale
  Pre-treatment SMQ | 20.0 (9.6) | 19.2 (9.5)
  Post-treatment SMQ | 26.2 (9.6) | 23.4 (9.5)
  6 month follow-up SMQ | 30.2 (11.9) | 27.6 (10.1)

6. Secondary Outcome: The Preschool Anxiety Scale - Parent Report
Description: The Preschool Anxiety Scale - Parent report (PAS-P) is a 29-item parent-report questionnaire for use with 3- to 6-year-old children. Parents report on their child's anxiety symptoms in different scenarios. Parents rate items on a 5-point Likert scale.
Time Frame: The PAS-P was completed by parents at all 3 time-points: 1) Pre-treatment (baseline), 2) Post-treatment, and 3) 6-month follow-up (from baseline date).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Taming Sneaky Fears Group | Parent Psychoeducation and Child Socialization Group
Number analyzed (Participants) | 46 | 44
units on a scale
  Pre-treatment PAS-P Score | 36.7 (20.2) | 39.6 (16.3)
  Post-treatment PAS-P Score | 32.3 (16) | 35.8 (13.4)
  6 month follow-up PAS-P Score | 26.5 (16) | 31.4 (17.5)

ADVERSE EVENTS:
Time Frame: Adverse events were assessed from September 2015 - December 2017, from treatment start date, to 6 months following administration. Adverse events were collected through self-report and participants were encouraged to share any concerns. However, given that this was a psychotherapy trial, no participants reported any adverse events.
Arm/Group | Taming Sneaky Fears Group | Parent Psychoeducation and Child Socialization Group
All-Cause Mortality (participants affected / at risk) | 0/46 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/44
Other Adverse Events (participants affected / at risk) | 0/46 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT02554929/Prot_SAP_000.pdf